CLINICAL TRIAL: NCT03221517
Title: Mapping the Shift Worker's Microbiome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carsten Skarke, MD, Research Assistant Professor, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 826117
Record Dates: First submitted 2016-12-21; First posted 2017-07-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Shift workers receive a standardized meal with a glucose challenge test
  Interventions: Other: Standardized meal with a glucose challenge test
- Cohort 2 (Experimental): Matched healthy controls receive a standardized meal with a glucose challenge test
  Interventions: Other: Standardized meal with a glucose challenge test

INTERVENTIONS:
Other: Standardized meal with a glucose challenge test — Postprandial glucose and insulin response

SUMMARY:
The investigators hypothesize that disruptions to the microbiome of shift-workers represent a hitherto unexamined factor contributing to disease risk. The investigators will therefore define time-of-day dependent fluctuations of the microbiome in night shift workers and matched daytime workers deeply phenotyped for behavioral, clinical, and metabolomic outputs using integrated remote sensing.

DETAILED DESCRIPTION:
Though several epidemiological studies have demonstrated that working night shift schedules are a risk factor for developing metabolic and cardiovascular diseases, the mechanisms through which this is conferred is not yet understood. Shift-work schedules alter employee's patterns of activity, light exposure and dietary intake in a manner incongruent with the endogenous clock. This circadian clock ensures that our metabolic activity occurs at maximally beneficial times of the day, but is largely unable to adapt to rapidly shifting schedules or sustained night-work. In mice, the investigators' lab has previously shown that genes relevant to all aspects of the metabolic syndrome are subject to circadian oscillation and that the gut microbiome is also subject to control by the host molecular clock. Despite the large contribution of our microbiome to host metabolism, the microbiome has been scarcely studied in the shift-working population. The investigators hypothesize that disruptions to the microbiome of shift-workers represent a hitherto unexamined factor contributing to disease risk. The investigators will therefore define time-of-day dependent fluctuations of the microbiome in night shift workers and matched daytime workers deeply phenotyped for behavioral, clinical, and metabolomic outputs using integrated remote sensing. The investigators will assess core body temperature, sleep/activity cycles, cortisol and melatonin as outputs determined by the host clock, and postprandial glucose and insulin levels as well as nocturnal blood pressure dipping as risk-related outputs. Through antibiotic-induced suppression, The investigators will determine the microbiome's specific contribution to these outputs. This has major implications for refining shift-work schedules and exploring therapeutic strategies in this population.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: healthy un-medicated males (to limit gender-induced variability similar to our pilot study), shift-work schedule (>3 shifts per month outside 7am-6pm (9)) for the past ≥10 years, 40-59 years old (increased prevalence of the metabolic syndrome at ≥60 years of age (20));
* Cohort 2: day workers who work 7am-6pm for ≥10 years matched for line of work, age, gender, and BMI;
* Volunteers are capable of giving informed consent;
* 40-59 years of age;
* Own an android smartphone which installs the remote sensing applications (those with apple smartphones will not be recruited);
* Non-smoking;
* Male subjects
* The use of contraception will NOT be required for male participants.

Exclusion Criteria:

* Recent travel across more than two (2) time zones (within the past month);
* Planned travel across more than two (2) time zones during the planned study activities;
* Use of illicit drugs;
* High dose vitamins (Vitamin A, Vitamin C, Vitamin E, Beta Carotene, Folic Acid and Selenium), alcohol and any over-the counter NSAID in the (2) two weeks before the start of the 48 hour deep phenotyping;
* High fat foods and caffeine in the past 24 hours prior to the 48-hour deep chronotyping session;
* History of abdominal surgery;
* Known allergy or intolerance to Vancomycin, and/or Neomycin;
* Use of anticholinergics in the week prior to the 48-hour sessions;
* Use of laxatives or anti-diarrhea medications in the two weeks prior to the 48-hour sessions;
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening;
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject;

Ages: 40 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-09-27 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Area under the glucose over time curve | 12 hour
  Area under the curve (AUC) will be calculated from serial, timed glucose measurements

SECONDARY OUTCOMES:
Time-of-day dependent fluctuations of the microbiome | 48 hours
  Relative abundances assessed several times of day (morning, afternoon, evening, night with target times of 08:00, 14:00, 20:00, 02:00 +/- 1 hour)
Compound outcome derived from percent variance explained in communication (number of phone calls and text messages), mobility (miles traveled), light exposure, blood pressure, heart rate, heart rate variability, sleep/wake times, body core temperature | 48 hours
  To evaluate the linear relationships between every pairwise combination of variables in the integrated dataset, the R^2, or coefficient of determination, will be calculated for each pair using linear regression. A heat map of the proportion of variance in each variable (e.g. mobility, light exposure, systolic blood pressure) explained by each other variable will then be constructed to allow an integrative exploration of these data. Here, the advantage is that multiple assessments with different units of measure can be integrated to generate deep phenotypes.
Compound outcome derived from variance observed in multiomics outputs (metabolites, microbiota). | 48 hours
  To explore factors contributing to the variance observed using principal components analysis

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skarke, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No